CLINICAL TRIAL: NCT03436628
Title: Using an mHealth App to Transition Care of Type-1 Diabetes From Parents to Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Sparrow Health System (Other)
Responsible Party: Principal Investigator, Bree Holtz, Assistant Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MyT1DHero
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes Mellitus; Adolescent Behavior; Parent-Child Relations; Communication
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Adolescent Behavior; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App Use (Experimental): Kids (10-15 years old) with type 1 diabetes and one of their parents will receive the MyT1DHero app to use for a 3-month period. Participants are urged to use the app four times each day.
  Interventions: Device: MyT1DHero

INTERVENTIONS:
Device: MyT1DHero — A mobile phone application

SUMMARY:
Type 1 diabetes (T1D) afflicts approximately 154,000 people under the age of 20. Most people with T1D are diagnosed at a young age; their parents have to manage their child's condition. Eventually, the child must begin to take steps to transition to self-management. During the transition from parent to adolescent self-management, difficulties arise because adolescents may not be fully aware of, or want, to take responsibility for all the necessary tasks to successfully manage their T1D. Though there are other apps on the market to help with diabetes care, NONE do what the proposed app will do. The proposed self-management mobile app allows for monitoring the patients' T1D by linking their self-management information to their parents' cell phone, and thus also helps to bridge communication gaps. Prior research suggests that these are critical gaps that must be filled in order for successful transition in care to occur, the proposed app will help fill some of these gaps.

ELIGIBILITY:
Inclusion Criteria:

The adolescents must:

1. have a T1D diagnosis according to the ADA practice guidelines;
2. be 10 to 15 years old;
3. have had a diagnosis of T1D for at least six months;
4. have an A1c > 7;97
5. have had at least two outpatient visits in the past two years;
6. be treated at Sparrow for diabetes;
7. be fluent in English;
8. have a parent/guardian willing to participate;
9. be allowed to use a mobile phone for the study;
10. have permission from their care team.

The parent/guardian must:

1. have an adolescent with T1D who is 10 to 15 years old;
2. be fluent in English;
3. have daily access to email and the Internet (for appointment reminders and technical support).

Exclusion Criteria:

The exclusions for adolescents include:

1. significant medical conditions other than T1D;
2. being treated for thyroid disorders, celiac disease, or eating disorders;
3. being in foster care.

Exclusion criteria for both the adolescents and parents/guardians include:

a) a diagnosis of a major psychiatric or neurocognitive disorder (e.g., traumatic brain injury, dementia, schizophrenia, bipolar disorder, borderline personality disorder, and mental retardation).

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to Self-management | Baseline and 3 months
  Measured with the Diabetes Behavior Rating Scale (5 point likert scale, never-always); A higher value represents a better outcome
Change in Hemoglobin A1c (HbA1c) | Baseline and 3 months
  A laboratory test of HbA1c will be collected at the local hospital; A lower value represents a better outcome

SECONDARY OUTCOMES:
Change in Social Support | Baseline and 3 months
  Measured with the Multidimensional Scale of Perceived Social Support (5 point likert scale, all of the time-never); A lower value represents a better outcome
Change in Self-Efficacy | Baseline and 3 months
  Measured using Diabetes Empowerment Scale - Short Form (5-point likert scale, strongly disagree-strongly agree); A higher value represents a better outcome
Change in Quality of Life | Baseline and 3 months
  Measured using PedsQL (5-point likert scale, never-almost always); A higher value represents a better outcome
Change in Conflict | Baseline and 3 months
  Measured using Diabetes Family Conflict Scale (3-point likert scale, always-never); A lower value represents a better outcome
Parenting | Baseline
  Measured using Alabama Parenting Questionnaire (5-point likert scale, very often-never); Values of this scale vary based on which sub scale is being used. For negative parenting sub scales, a lower value represents a better outcome; and for positive parenting sub scales, a higher value represents a better outcome.
Change in Parental Monitoring | Baseline and 3 months
  Measured using Parental Monitoring of Diabetes Care Scale (5-point likert scale, always-never); A lower value represents a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bree M Holtz, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holtz B, Mitchell KM, Holmstrom AJ, Cotten SR, Dunneback JK, Jimenez-Vega J, Ellis DA, Wood MA. An mHealth-Based Intervention for Adolescents With Type 1 Diabetes and Their Parents: Pilot Feasibility and Efficacy Single-Arm Study. JMIR Mhealth Uhealth. 2021 Sep 14;9(9):e23916. doi: 10.2196/23916. PMID 34519670
- [Derived] Holtz BE, Mitchell KM, Hershey DD, Cotten SR, Holmstrom AJ, Richman J, Dunneback JK, Wood MA. Using an mHealth App to Transition Care of Type 1 Diabetes from Parents to Teens: Protocol for a Pilot Study. JMIR Res Protoc. 2018 Oct 30;7(10):e10803. doi: 10.2196/10803. PMID 30377142
- See also: Study Information Website — http://myt1d.org